CLINICAL TRIAL: NCT03505879
Title: Next Generation Sequencing to Detect Borrelia Burgdorferi DNA in the Blood of Pediatric Patients With Lyme Disease
Brief Title: Next Generation Sequencing Detection of Lyme Disease
Status: Completed | Type: Observational
Sponsor: Stony Brook University (Other)
Collaborators: Karius, Inc. (Industry)
Responsible Party: Principal Investigator, Christy Beneri, Assistant Professor of Pediatrics, Stony Brook University
Other Study IDs: 1205731-1
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Lyme Disease; Pediatric Infectious Disease; Erythema Migrans; Lyme Arthritis; Lyme Carditis; Lyme Disease Meningitis
Keywords: Next Generation Sequencing
MeSH Terms: conditions — Lyme Disease; Glossitis, Benign Migratory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples for detection of infectious pathogens by next generation sequencing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Next Generation Sequencing is capable of sequencing millions of small strands of DNA from a single blood sample, potentially improving its sensitivity compared to PCR testing, which only detects predetermined larger strands of DNA. We will test the ability of NGS to detect Borrelia burgdorferi DNA in the blood of pediatric patients with Lyme disease. We will conduct an observational study of NGS testing on pediatric patients at all stages of Lyme disease. Study involvement will require a single study visit for clinical data collection and blood draw. We will enroll patients at all phases of suspected Lyme disease, collect clinically relevant information, and test for Lyme disease using Next Generation Sequencing and standard Lyme serologic testing. If the patient has multiple erythema migrans, Lyme meningitis, facial nerve palsy, arthritis, or carditis, a B. burgdorferi serum PCR will also be sent. Enrollment and Next Generation Sequencing blood draw will occur before or up to 24 hours after the first dose of antibiotics is administered. We will also study the impact of antibiotics on NGS testing by running the test 6-24 hours after antibiotics are started among a small subset of patients with a multiple erythema migrans rash. Collected data will be analyzed with basic descriptive statistics.

ELIGIBILITY:
Lyme disease subjects (Cases):

Inclusion criteria:

1. Age 1 to <18 years old
2. The subject has spent time in a Lyme-endemic area during the previous month
3. The subject has a suspected Lyme disease infection

Exclusion criteria:

1. Past infection with Lyme disease
2. Received oral or IV antibiotics within 1 month prior to presentation Note: Subjects may be enrolled if NGS blood test can be drawn <24 hours after the first dose of Lyme diseasetargeted antibiotics is administered

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cases will include pediatric patients age 1 to <18 years old who currently have a specific Lyme disease syndrome and have been on antibiotics for less than 24 hours prior to blood draw
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Ability of Next Generation Sequencing to detect Borrelia burgdorferi DNA in blood | 1 year
  To determine if Next Generation Sequencing (NGS) is able to detect Borrelia burgdorferi DNA in the blood of pediatric patients with Lyme disease, including those with erythema migrans (single or multiple), Lyme meningitis, Lyme carditis, Lyme disease facial palsy, and Lyme arthritis
NGS detection of Borrelia burgdorferi DNA following antibiotics | 1 year
  To determine if Next Generation Sequencing (NGS) is able to detect Borrelia burgdorferi DNA in the blood of pediatric patients with a multiple erythema migrans rash shortly after the first dose of antibiotics.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Setauket, New York, United States

REFERENCES:
- [Background] Schwartz AM, Hinckley AF, Mead PS, Hook SA, Kugeler KJ. Surveillance for Lyme Disease - United States, 2008-2015. MMWR Surveill Summ. 2017 Nov 10;66(22):1-12. doi: 10.15585/mmwr.ss6622a1. PMID 29120995
- [Background] Theel ES. The Past, Present, and (Possible) Future of Serologic Testing for Lyme Disease. J Clin Microbiol. 2016 May;54(5):1191-6. doi: 10.1128/JCM.03394-15. Epub 2016 Feb 10. PMID 26865690
- [Background] Aguero-Rosenfeld ME, Wang G, Schwartz I, Wormser GP. Diagnosis of lyme borreliosis. Clin Microbiol Rev. 2005 Jul;18(3):484-509. doi: 10.1128/CMR.18.3.484-509.2005. PMID 16020686
- [Background] Babady NE, Sloan LM, Vetter EA, Patel R, Binnicker MJ. Percent positive rate of Lyme real-time polymerase chain reaction in blood, cerebrospinal fluid, synovial fluid, and tissue. Diagn Microbiol Infect Dis. 2008 Dec;62(4):464-6. doi: 10.1016/j.diagmicrobio.2008.08.016. Epub 2008 Oct 22. PMID 18947959
- [Background] Kalish RA, McHugh G, Granquist J, Shea B, Ruthazer R, Steere AC. Persistence of immunoglobulin M or immunoglobulin G antibody responses to Borrelia burgdorferi 10-20 years after active Lyme disease. Clin Infect Dis. 2001 Sep 15;33(6):780-5. doi: 10.1086/322669. Epub 2001 Aug 10. PMID 11512082
- [Background] da Fonseca AJ, Galvao RS, Miranda AE, Ferreira LC, Chen Z. Comparison of three human papillomavirus DNA detection methods: Next generation sequencing, multiplex-PCR and nested-PCR followed by Sanger based sequencing. J Med Virol. 2016 May;88(5):888-94. doi: 10.1002/jmv.24413. Epub 2015 Nov 6. PMID 26496186
- [Background] Abril MK, Barnett AS, Wegermann K, Fountain E, Strand A, Heyman BM, Blough BA, Swaminathan AC, Sharma-Kuinkel B, Ruffin F, Alexander BD, McCall CM, Costa SF, Arcasoy MO, Hong DK, Blauwkamp TA, Kertesz M, Fowler VG Jr, Kraft BD. Diagnosis of Capnocytophaga canimorsus Sepsis by Whole-Genome Next-Generation Sequencing. Open Forum Infect Dis. 2016 Jul 12;3(3):ofw144. doi: 10.1093/ofid/ofw144. eCollection 2016 Sep. PMID 27704003